CLINICAL TRIAL: NCT00110604
Title: The Folic Acid and Carotid Intima-Media Thickness (FACIT) Study: A Randomized Controlled Trial
Brief Title: The Effect of Folic Acid on Atherosclerosis, Cognitive Performance and Hearing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Wageningen Centre for Food Sciences (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pou.0224L; ZonMw 20010002
Record Dates: First submitted 2005-05-10; First posted 2005-05-11 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2005-05

CONDITIONS: Atherosclerosis; Vascular Disease; Cognitive Decline; Hearing Loss; Inflammation; Age-Related Memory Disorder
Keywords: Folic acid; Atherosclerosis; Cognitive function; Hearing; Inflammation; Hemostasis; Arterial stiffness
MeSH Terms: conditions — Atherosclerosis; Vascular Diseases; Cognitive Dysfunction; Hearing Loss; Inflammation; Memory Disorders | interventions — Folic Acid

INTERVENTIONS:
Behavioral: folic acid (0.8 mg)

SUMMARY:
The purpose of this study is to determine if folic acid supplementation can slow down atherosclerotic progression, age-related cognitive decline and age-related hearing loss.

DETAILED DESCRIPTION:
Low levels of B vitamins, in particular folate, and high levels of plasma total homocysteine, have been associated with a variety of age-related diseases and disorders, including cardiovascular disease, dementia and hearing impairment. Extra folate, for example in the form of folic acid, is known to decrease the concentrations of plasma total homocysteine.

We examined whether 0.8 mg/d folic acid could slow down atherosclerotic progression and the above mentioned age-related processes.

ELIGIBILITY:
Inclusion Criteria:

* 50-70 years
* Men and post-menopausal women
* Women with a surgically removed uterus were required to be >=55 years

Exclusion Criteria:

* Plasma total homocysteine <13 or >26 umol/L
* Serum vitamin B12 <200 pmol/L
* Self-reported current use of drugs which affect folate metabolism
* Self-reported current use of drugs believed to influence intima-media thickening, i.e., lipid-lowering drugs, hormone replacement therapy
* Self-reported medical diagnosis of renal, intestinal, thyroid disease
* Self-reported medical diagnosis of current cancer
* Self-reported current use of supplements containing B vitamins
* Self-reported inability or unwillingness to fast for 12 hours
* <80% compliance using placebo pills during a 6-week run-in period
* Not giving written informed consent
* Participation in other research studies

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 835
Dates: Start 2000-09; Study Completion 2004-12

PRIMARY OUTCOMES:
Change in mean carotid intima-media thickness
Change in maximum carotid intima-media thickness

SECONDARY OUTCOMES:
Change in carotid distension
Change in hearing levels (pure tone air conduction averages of 0.5, 1, and 2 kHz & 4, 6 and 8 kHz)
Cognitive performance at year 3 (cognitive domains: simple speed, cognitive flexibility, and memory; and information processing speed and semantic memory)
Inflammatory markers and hemostasis markers

CONTACTS AND LOCATIONS:
Overall Officials: Petra Verhoef, PhD, Principal Investigator — Wageningen Centre for Food Sciences
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] van Soest APM, van de Rest O, Witkamp RF, de Groot LCPGM. Positive effects of folic acid supplementation on cognitive aging are dependent on omega-3 fatty acid status: a post hoc analysis of the FACIT trial. Am J Clin Nutr. 2021 Apr 6;113(4):801-809. doi: 10.1093/ajcn/nqaa373. PMID 33564824
- [Derived] Jung AY, Smulders Y, Verhoef P, Kok FJ, Blom H, Kok RM, Kampman E, Durga J. No effect of folic acid supplementation on global DNA methylation in men and women with moderately elevated homocysteine. PLoS One. 2011;6(9):e24976. doi: 10.1371/journal.pone.0024976. Epub 2011 Sep 23. PMID 21966393
- [Derived] Schiepers OJ, van Boxtel MP, de Groot RH, Jolles J, Kok FJ, Verhoef P, Durga J. DNA methylation and cognitive functioning in healthy older adults. Br J Nutr. 2012 Mar;107(5):744-8. doi: 10.1017/S0007114511003576. Epub 2011 Jul 27. PMID 21791146
- [Derived] Durga J, Bots ML, Schouten EG, Grobbee DE, Kok FJ, Verhoef P. Effect of 3 y of folic acid supplementation on the progression of carotid intima-media thickness and carotid arterial stiffness in older adults. Am J Clin Nutr. 2011 May;93(5):941-9. doi: 10.3945/ajcn.110.006429. Epub 2011 Mar 23. PMID 21430116
- [Derived] Durga J, van Boxtel MP, Schouten EG, Kok FJ, Jolles J, Katan MB, Verhoef P. Effect of 3-year folic acid supplementation on cognitive function in older adults in the FACIT trial: a randomised, double blind, controlled trial. Lancet. 2007 Jan 20;369(9557):208-16. doi: 10.1016/S0140-6736(07)60109-3. PMID 17240287
- [Derived] Durga J, Verhoef P, Anteunis LJ, Schouten E, Kok FJ. Effects of folic acid supplementation on hearing in older adults: a randomized, controlled trial. Ann Intern Med. 2007 Jan 2;146(1):1-9. doi: 10.7326/0003-4819-146-1-200701020-00003. PMID 17200216
- See also: FACIT study website — http://www.theheart.org/article/765625.do